CLINICAL TRIAL: NCT07096089
Title: Effect of Whole-body Vibration on Shoulder Proximal Stability in Children With Cerebral Palsy
Brief Title: Effect of Vibration on Shoulder Proximal Stability in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Usama Mahmoud Ahmed, Lecturer at Department of Physical Therapy for Paediatrics, Faculty of Physical Therapy, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004848
Record Dates: First submitted 2025-07-21; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Proximal stability; Shoulder; Whole body vibration
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Experimental trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional physical therapy program and Sling exercise therapy (Experimental): Conventional physical therapy program and Sling exercise therapy
  Interventions: Procedure: Conventional physical therapy program and Sling exercise therapy
- Whole body vibration (Experimental): Whole body vibration
  Interventions: Procedure: Whole body vibration

INTERVENTIONS:
Procedure: Conventional physical therapy program and Sling exercise therapy — The control group received a conventional physical therapy program in addition to sling exercise therapy (SET) for 60 minutes.
  Arms: Conventional physical therapy program and Sling exercise therapy
Procedure: Whole body vibration — The study group received the same selected conventional physical therapy program in addition to sling exercise therapy (SET) given to the control group (for 30 minutes) besides whole body vibration (WBV) (for 30 minutes).
  Arms: Whole body vibration

SUMMARY:
Objectives: Children with cerebral palsy have weak proximal stability which not only affects range of available motion but also reflects on distal dexterity. These have a great impact on their mobility and efficiency of daily living activities. Vibration has been regarded as an effective exercise method to improve muscle strength and endurance. The aim of this study was to determine the effect of vibration on shoulder proximal stability in children with cerebral palsy.

Methods: Fifty children with cerebral palsy from 4 to 9 years old participated in this study and were selected from the outpatient clinic of faculty of physical therapy. They were divided into two groups of equal sizes randomly. The control group received a conventional physical therapy program in addition to Sling exercise therapy, and the study group received the same conventional physical therapy program in addition to Sling exercise therapy (SET) and Whole-body vibration (WBV). Shoulder muscle strength was assessed for both groups by using Lafayette manual muscle tester before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* children with cerebral palsy affecting weight bearing of the upper limbs.
* Aged from 4 to 9 years.
* Both gender participated.
* Having grade 1 and 1+ spasticity according to the Modified Ashworth Scale.

Exclusion Criteria:

* Congenital anomalies.
* Surgical or neurological disease of the upper limbs.
* Osteopenia or osteoporosis.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Shoulder muscle strength | 4 to 6 months
  Lafayette manual muscle tester In order to produce precise, objective, and dependable findings, the Lafayette Manual Muscle Tester (MMT) Model Number 01163 blends modern ergonomic design with accuracy and precision. The three cushioned stirrups that were interchangeable allowed for the confident and efficient use of recognized techniques while maintaining patient comfort.
  No other manual muscle test method uses the advancements found in the Lafayette MMT. The user may choose from an extensive array of variables through the interactive menus, including high and low threshold settings (to account for larger muscles or fingers), test periods ranging from one to ten seconds, and data storage. There is less chance of reading mistakes or selecting undesirable alternatives because of the wide, easy-to-read LCD screen that clearly shows all the information.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical therapy, Cairo University, Giza, Office Post Cairo University Giza, Egypt

IPD SHARING:
Plan to Share IPD: No